CLINICAL TRIAL: NCT07153276
Title: TREATMENT OF VAGINAL DRYNESS IN SJÖGREN'S DISEASE WITH CO2-LASER VERSUS TOPICAL PROMESTRIENE: A PROSPECTIVE RANDOMIZED STUDY
Brief Title: TREATMENT OF VAGINAL DRYNESS IN SJÖGREN'S DISEASE WITH CO2-LASER VERSUS TOPICAL PROMESTRIENE
Acronym: VaLS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67377523.3.0000.0068
Record Dates: First submitted 2025-08-20; First posted 2025-09-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sjogren Syndrome; Sjogren Disease; Primary Sjogren Syndrome
Keywords: Sjogren syndrome; vaginal dryness; vaginitis sicca; vaginal fractional CO2 laser; promestriene
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SjD with sicca vagintis complaints treated with vaginal fractional CO2 laser (Experimental): Thirty SjD patients with vaginitis sicca symptoms allocated to the intervention group (vaginal fractional CO2 laser)
  Interventions: Device: Fractional CO2 laser (vaginal)
- SjD with sicca vagintis complaints treated with topical promestriene (Active Comparator): Thirty SjD patients with vaginitis sicca symptoms allocated to the comparator group (topical promestriene)
  Interventions: Drug: Promestriene Vaginal

INTERVENTIONS:
Device: Fractional CO2 laser (vaginal) — Vaginal fractional CO2 laser applications will be performed once a month for three consecutive months.
  Arms: SjD with sicca vagintis complaints treated with vaginal fractional CO2 laser
Drug: Promestriene Vaginal — Patients in the group treated with promestriene will apply a 10 mg vaginal capsule at night for fifteen consecutive days and, after this period, one application every three days, until completing six months of treatment.
  Arms: SjD with sicca vagintis complaints treated with topical promestriene

SUMMARY:
Sjögren's disease (SjD) is a chronic, immune-mediated, systemic inflammatory disease characterized mainly by involvement of the salivary and lacrimal glands, causing symptoms of sicca syndrome. The disease predominantly affects women (9:1 to 20:1), with a peak incidence between 40 and 60 years of age. Symptoms of dryness include those resulting from vaginitis sicca, such as vulvovaginal irritation, dryness, pruritus, dyspareunia, polyuria, nocturia, dysuria, and urinary urgency/incontinence, which may begin before and worsen after menopause. These symptoms impact the sexual life and health-related quality of life of SjD patients. However, there are no specific recommendations for the management of vaginal dryness in this disease. Urogenital syndrome (UGS), a condition that affects women from the general population in the menopausal phase, is characterized by similar symptoms and can be treated with systemic or local hormone therapy (e.g., topical promestriene). Current data also demonstrate the efficacy and safety of vaginal fractional CO2 laser treatment for UGS. However, there are no studies on the efficacy of vaginal fractional CO2 laser and topical promestriene in the treatment of vaginal dryness in SjD.

DETAILED DESCRIPTION:
This is a prospective randomized study lasting 6 months. Sixty SjD patients (pre- or post-menopausal) and with complaints of vaginal dryness will be included and randomized into two groups: 30 patients for the intervention group - vaginal fractional CO2 laser - and 30 patients for the comparator group - topical promestriene. Vaginal fractional CO2 laser applications will be performed once a month for three consecutive months. Patients in the group treated with promestriene will apply a 10 mg vaginal capsule at night for fifteen consecutive days and, after this period, one application every three days, until completing six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SjD according to the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria (2016).
* Controlled systemic disease activity [EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI)] < 5 and without use of glucocorticoids or with a maximum dose of prednisone of 15 mg/day.
* Present complaints of vaginal dryness upon study entry.
* Agreeing to participate in the protocol according to the informed consent form signed before study inclusion.

Exclusion Criteria:

* History of breast, uterine or ovarian neoplasia, history of thromboembolic events, heart, kidney or liver failure.
* Other associated autoimmune rheumatic diseases, such as spondyloarthritis, rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, dermatomyositis and mixed connective tissue disease.
* Conditions that may mimic SjD, such as history of head and neck radiation therapy, acquired immunodeficiency syndrome, hepatitis B and C, sarcoidosis, IgG4-related disease, and graft-versus-host disease.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2029-08-20 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Vaginal Health Index (VHI) | Four and six months
  To assess the improvement in the Vaginal Health Index (VHI) after treatment compared to the patient's baseline status in both arms. This score ranges from 5 (minimum) to 25 (maximum) and higher values indicate better outcomes.

SECONDARY OUTCOMES:
6-Item version of the Female Sexual Function Index (FSFI) | Four and six months
  To assess the improvement in the 6-item version of the Female Sexual Function Index (FSFI) after treatment compared to the patient's baseline status in both arms. This score ranges from 0 (minimum) to 30 (maximum) and higher values indicate better outcomes.
Primary Sjögren's Syndrome Quality of Life questionnaire (PSSQoL) | Four and six months
  To assess the improvement in the Primary Sjögren's Syndrome Quality of Life questionnaire (PSSQoL) after treatment compared to the patient's baseline status in both arms. This score ranges from 0 (minimum) to 96 (maximum) and higher values indicate worse outcomes.
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | Four and six months
  To assess the improvement in the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) after treatment compared to the patient's baseline status in both arms. This score ranges from 0 (minimum) to 21 (maximum) and higher values indicate worse outcomes.
Visual analogue scale (VAS) of vaginal dryness symptoms | Four and six months
  To assess the improvement in the visual analogue scale (VAS) of vaginal dryness symptoms after treatment compared to the patient's baseline status in both arms. This scale ranges from 0 (minimum) to 10 (maximum) and higher values indicate worse outcomes.
Persistence of the beneficial effects of laser therapy - visual analogue scale (VAS) of vaginal dryness symptoms | Six months
  To assess the possible persistence of the beneficial effects of laser therapy after the end of applications (in the medium term). This assessment will be performed by observing improvements on the visual analogue scale (VAS) of vaginal dryness symptoms after treatment compared to the patient's baseline status in both arms. This scale ranges from 0 (minimum) to 10 (maximum) and higher values indicate worse outcomes.
Incidence of treatment-emergent adverse events (safety and tolerability) | One month, two months, three months, four months, five months, six months
  To assess the incidence of treatment-emergent adverse events (as a percentage) in the two arms of the study.
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) (safety and tolerability) | Four and six months
  To assess the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) after treatment compared to the patient's baseline status in both study arms. This score ranges from 0 (minimum) to 123 (maximum) and higher values indicate worse outcomes.

OTHER OUTCOMES:
Histological analysis of vaginal wall biopsies before and after treatment | Six months
  To evaluate the improvement of histological parameters in the tissue samples from vaginal wall biopsies before and after treatment in the two arms of the study. An experienced pathologist will blindly evaluate the tissue samples from vaginal wall biopsies before and after interventions in both study arms. This pathologist will report their subjective assessment of improvement (increase) (yes or no) in epithelial thickness, collagen fibers (percentage of collagen types I and III), and/or microvascularization (weak, moderate and intense).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abstracts of the International Continence Society 31st annual meeting. Seoul, Korea, 18-21 September 2001. Neurourol Urodyn. 2001;20(4):371-576. No abstract available. PMID 11522151
- [Background] Tamanini JT, Dambros M, D'Ancona CA, Palma PC, Rodrigues Netto N Jr. [Validation of the "International Consultation on Incontinence Questionnaire -- Short Form" (ICIQ-SF) for Portuguese]. Rev Saude Publica. 2004 Jun;38(3):438-44. doi: 10.1590/s0034-89102004000300015. Epub 2004 Jul 8. Portuguese. PMID 15243675
- [Background] Dall'Agno ML, Ferreira CF, Ferreira FV, Perez-Lopez FR, Wender MCO. Validation of the Six-item Female Sexual Function Index in Middle-Aged Brazilian Women. Rev Bras Ginecol Obstet. 2019 Jul;41(7):432-439. doi: 10.1055/s-0039-1692694. Epub 2019 Jul 25. PMID 31344717
- [Background] Isidori AM, Pozza C, Esposito K, Giugliano D, Morano S, Vignozzi L, Corona G, Lenzi A, Jannini EA. Development and validation of a 6-item version of the female sexual function index (FSFI) as a diagnostic tool for female sexual dysfunction. J Sex Med. 2010 Mar;7(3):1139-46. doi: 10.1111/j.1743-6109.2009.01635.x. Epub 2009 Dec 1. PMID 19968774
- [Background] van Nimwegen JF, van der Tuuk K, Liefers SC, Verstappen GM, Visser A, Wijnsma RF, Vissink A, Hollema H, Mourits MJE, Bootsma H, Kroese FGM. Vaginal dryness in primary Sjogren's syndrome: a histopathological case-control study. Rheumatology (Oxford). 2020 Oct 1;59(10):2806-2815. doi: 10.1093/rheumatology/keaa017. PMID 32044981
- [Background] van Nimwegen JF, Arends S, van Zuiden GS, Vissink A, Kroese FG, Bootsma H. The impact of primary Sjogren's syndrome on female sexual function. Rheumatology (Oxford). 2015 Jul;54(7):1286-93. doi: 10.1093/rheumatology/keu522. Epub 2015 Feb 4. PMID 25652072
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome: A Consensus and Data-Driven Methodology Involving Three International Patient Cohorts. Arthritis Rheumatol. 2017 Jan;69(1):35-45. doi: 10.1002/art.39859. Epub 2016 Oct 26. PMID 27785888
- [Background] Serrano EV, Valim V, Miyamoto ST, Giovelli RA, Paganotti MA, Cade NV. Transcultural adaptation of the "EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI)" into Brazilian Portuguese. Rev Bras Reumatol. 2013 Nov-Dec;53(6):483-93. doi: 10.1016/j.rbr.2013.04.003. English, Portuguese. PMID 24477727
- [Background] Seror R, Ravaud P, Mariette X, Bootsma H, Theander E, Hansen A, Ramos-Casals M, Dorner T, Bombardieri S, Hachulla E, Brun JG, Kruize AA, Praprotnik S, Tomsic M, Gottenberg JE, Devauchelle V, Devita S, Vollenweider C, Mandl T, Tzioufas A, Carsons S, Saraux A, Sutcliffe N, Vitali C, Bowman SJ; EULAR Sjogren's Task Force. EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI): development of a consensus patient index for primary Sjogren's syndrome. Ann Rheum Dis. 2011 Jun;70(6):968-72. doi: 10.1136/ard.2010.143743. Epub 2011 Feb 22. PMID 21345815
- [Background] Seror R, Ravaud P, Bowman SJ, Baron G, Tzioufas A, Theander E, Gottenberg JE, Bootsma H, Mariette X, Vitali C; EULAR Sjogren's Task Force. EULAR Sjogren's syndrome disease activity index: development of a consensus systemic disease activity index for primary Sjogren's syndrome. Ann Rheum Dis. 2010 Jun;69(6):1103-9. doi: 10.1136/ard.2009.110619. Epub 2009 Jun 28. PMID 19561361
- [Background] Seganfredo IB, Bianchi C, Tacla M, Chedraui P, Haddad JM, Simoes R, Baracat EC, Soares JM Jr. Comparison of promestriene with vaginal fractional CO2 laser and radiofrequency treatments of genitourinary syndrome of menopause. Maturitas. 2024 Aug;186:108008. doi: 10.1016/j.maturitas.2024.108008. Epub 2024 Apr 24. PMID 38714422
- [Background] Samuels JB, Garcia MA. Treatment to External Labia and Vaginal Canal With CO2 Laser for Symptoms of Vulvovaginal Atrophy in Postmenopausal Women. Aesthet Surg J. 2019 Jan 1;39(1):83-93. doi: 10.1093/asj/sjy087. PMID 29726916
- [Background] Salvatore S, Ruffolo AF, Phillips C, Athanasiou S, Cardozo L, Serati M; EUGA Working Group. Vaginal laser therapy for GSM/VVA: where we stand now - a review by the EUGA Working Group on Laser. Climacteric. 2023 Aug;26(4):336-352. doi: 10.1080/13697137.2023.2225766. Epub 2023 Jul 3. PMID 37395104
- [Background] Priori R, Minniti A, Derme M, Antonazzo B, Brancatisano F, Ghirini S, Valesini G, Framarino-dei-Malatesta M. Quality of Sexual Life in Women with Primary Sjogren Syndrome. J Rheumatol. 2015 Aug;42(8):1427-31. doi: 10.3899/jrheum.141475. Epub 2015 Jul 1. PMID 26136488
- [Background] Politano CA, Costa-Paiva L, Aguiar LB, Machado HC, Baccaro LF. Fractional CO2 laser versus promestriene and lubricant in genitourinary syndrome of menopause: a randomized clinical trial. Menopause. 2019 Aug;26(8):833-840. doi: 10.1097/GME.0000000000001333. PMID 31246661
- [Background] Piccioni MG, Merlino L, Deroma M, Del Prete F, Tabacco S, Monti M, Benedetti Panici P. The impact of primary Sjogren's syndrome on female sexual function. Minerva Ginecol. 2020 Feb;72(1):50-54. doi: 10.23736/S0026-4784.20.04494-9. PMID 32153164
- [Background] Paganotti MA, Valim V, Serrano EV, Miyamoto ST, Giovelli RA, Santos MC. Validation and psychometric properties of the Eular Sjogren's Syndrome Patient Reported Index (ESSPRI) into Brazilian Portuguese. Rev Bras Reumatol. 2015 Sep-Oct;55(5):439-45. doi: 10.1016/j.rbr.2015.06.004. Epub 2015 Aug 6. English, Portuguese. PMID 26345467
- [Background] Miyamoto ST, Serrano EV, Gianordoli APE, Altoe LB, Noronha BD, Dos Santos PHA, Pedrini APT, da Silva NRS, Favarato LF, Alochio LV, Tome WA, Lackner A, Valim V. Brazilian version of the "Primary Sjogren's Syndrome - Quality of Life questionnaire (PSS-QoL)": translation, cross-cultural adaptation and validation. Adv Rheumatol. 2024 Aug 19;64(1):60. doi: 10.1186/s42358-024-00395-7. PMID 39160602
- [Background] Miyamoto ST, Paganotti MA, Serrano EV, Giovelli RA, Valim V. Assessment of fatigue and dryness in primary Sjogren's syndrome: Brazilian version of "Profile of Fatigue and Discomfort - Sicca Symptoms Inventory (short form) (PROFAD-SSI-SF)". Rev Bras Reumatol. 2015 Mar-Apr;55(2):113-22. doi: 10.1016/j.rbr.2014.10.002. Epub 2014 Nov 7. PMID 25582994
- [Background] Lackner A, Stradner MH, Hermann J, Unger J, Stamm T, Graninger WB, Dejaco C. Assessing health-related quality of life in primary Sjogren's syndrome-The PSS-QoL. Semin Arthritis Rheum. 2018 Aug;48(1):105-110. doi: 10.1016/j.semarthrit.2017.11.007. Epub 2017 Nov 27. PMID 29395257
- [Background] Isik H, Isik M, Aynioglu O, Karcaaltincaba D, Sahbaz A, Beyazcicek T, Harma MI, Demircan N. Are the women with Sjogren's Syndrome satisfied with their sexual activity? Rev Bras Reumatol Engl Ed. 2017 May-Jun;57(3):210-216. doi: 10.1016/j.rbre.2017.01.002. Epub 2017 Feb 8. English, Portuguese. PMID 28535892
- [Background] Haga HJ, Gjesdal CG, Irgens LM, Ostensen M. Reproduction and gynaecological manifestations in women with primary Sjogren's syndrome: a case-control study. Scand J Rheumatol. 2005;34(1):45-8. doi: 10.1080/03009740510017959. PMID 15903025
- [Background] Gozukucuk M, Turkyilmaz E, Kucuksahin O, Erten S, Ustun Y, Yavuz AF. Effects of primary Sjogren's syndrome on female genitalia and sexual functions. Clin Exp Rheumatol. 2021 Nov-Dec;39 Suppl 133(6):66-72. doi: 10.55563/clinexprheumatol/spnjy5. Epub 2021 Oct 6. PMID 34665702
- [Background] Filippini M, Porcari I, Ruffolo AF, Casiraghi A, Farinelli M, Uccella S, Franchi M, Candiani M, Salvatore S. CO2-Laser therapy and Genitourinary Syndrome of Menopause: A Systematic Review and Meta-Analysis. J Sex Med. 2022 Mar;19(3):452-470. doi: 10.1016/j.jsxm.2021.12.010. Epub 2022 Jan 29. PMID 35101378
- [Background] Farenhorst CA, de Wolff L, Arends S, van Nimwegen JF, Kroese FGM, Verstappen GM, Bootsma H. Clinical determinants of vaginal dryness in patients with primary Sjogren's syndrome. Clin Exp Rheumatol. 2021 Nov-Dec;39 Suppl 133(6):73-79. doi: 10.55563/clinexprheumatol/hzveng. Epub 2021 Oct 7. PMID 34665706
- [Background] Bowman SJ, Hamburger J, Richards A, Barry RJ, Rauz S. Patient-reported outcomes in primary Sjogren's syndrome: comparison of the long and short versions of the Profile of Fatigue and Discomfort--Sicca Symptoms Inventory. Rheumatology (Oxford). 2009 Feb;48(2):140-3. doi: 10.1093/rheumatology/ken426. Epub 2008 Dec 11. PMID 19074185
- [Background] Alvisi S, Gava G, Orsili I, Giacomelli G, Baldassarre M, Seracchioli R, Meriggiola MC. Vaginal Health in Menopausal Women. Medicina (Kaunas). 2019 Sep 20;55(10):615. doi: 10.3390/medicina55100615. PMID 31547180
- [Background] Aguiar LB, Politano CA, Costa-Paiva L, Juliato CRT. Efficacy of Fractional CO2 Laser, Promestriene, and Vaginal Lubricant in the Treatment of Urinary Symptoms in Postmenopausal Women: A Randomized Clinical Trial. Lasers Surg Med. 2020 Oct;52(8):713-720. doi: 10.1002/lsm.23220. Epub 2020 Jan 28. PMID 31990089